CLINICAL TRIAL: NCT02085291
Title: The Effect of Fluids and Norepinephrine for Mean Arterial Pressure Titration to Patients' Usual Levels on the Microcirculation of Initial Resuscitated Hypertensive Septic Shock Patients.
Brief Title: Effect of Different Strategies for Titrating a High MAP on Microcirculation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Zhongda Hospital, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014ZDll.2; Targeting microcirculation (Other: Zhongda Hospital)
Record Dates: First submitted 2014-02-28; First posted 2014-03-12 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Septic Shock; Hypertension
Keywords: septic shock; microcirculation; norepinephrine
MeSH Terms: conditions — Shock, Septic; Hypertension | interventions — Norepinephrine; Crystalloid Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resp-FL (Experimental): Patients received 500 ml crystalloid for fluid challenge within 20 minutes, then a PLR test was performed to predict fluid responsiveness. If the patient was fluid responsive, more 500 ml crystalloids were given until fluid nonresponsive. If the MAP still not achieved the target value, NE was increased to achieve the target one. The target MAP was maintain MAP within 10% of the reference value.
  Interventions: Drug: Crystalloid
- Resp-NE (Experimental): In Resp-NE group, norepinephrine was increased to enhance MAP within 10% of the reference value.
  Interventions: Drug: Norepinephrine
- Nonresp-NE (Experimental): In Nonresp-NE group, norepinephrine was increased to enhance MAP within 10% of the reference value.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine infusion to titrate MAP to usual level
  Other Names: NE group
  Arms: Nonresp-NE; Resp-NE
Drug: Crystalloid — Patients received 500 ml crystalloid for fluid challenge within 20 minutes, then a PLR test was performed to predict fluid responsiveness. If the patient was fluid responsive, more 500 ml crystalloids were given until fluid nonresponsive. If the MAP still not achieved the target value, NE was increased to achieve the target one.
  Other Names: Fluid group
  Arms: Resp-FL

SUMMARY:
Assess the effect of fluids and norepinephrine for mean arterial pressure titration to patients' usual level on the microcirculation of initial resuscitated hypertensive septic shock patients.

DETAILED DESCRIPTION:
Microcirculatory dysfunction plays an important role in the development of organ failure in patients with septic shock. Numerous studies focus on the effect of mean arterial pressure (MAP) titration on microcirculation, however, by what strategy is better for microcirculation in septic shock patients with previous hypertension is still a matter of debate. The goal of this study was to assess the effect of different strategies for MAP titration to individualized level on microcirculation in hypertensive septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

1. Hypertensive patients with septic shock for less than 24 hours. Septic shock was defined by the 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference.
2. Initial fluid resuscitation was performed to maintain the central venous pressure (CVP) for more than 8 mm Hg and central venous hemoglobin saturation for more than 70%.
3. Patients were still requiring NE to maintain the MAP of 65 mm Hg.

Exclusion Criteria:

1. had severe untreated or uncontrolled hypertension (systolic blood pressure more than 180 mm Hg or/and diastolic blood pressure more than 110 mm Hg);
2. were younger than 18 years old or pregnant;
3. were unable to acquire the usual level or resting level of blood pressure;
4. refused to participate the trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Perfused vessel density | 20 minutes
  Perfused vessel density of small vessels

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, Principal Investigator — Southeastt University
Locations (1):
- Nanjing Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rhee C, Dantes R, Epstein L, Murphy DJ, Seymour CW, Iwashyna TJ, Kadri SS, Angus DC, Danner RL, Fiore AE, Jernigan JA, Martin GS, Septimus E, Warren DK, Karcz A, Chan C, Menchaca JT, Wang R, Gruber S, Klompas M; CDC Prevention Epicenter Program. Incidence and Trends of Sepsis in US Hospitals Using Clinical vs Claims Data, 2009-2014. JAMA. 2017 Oct 3;318(13):1241-1249. doi: 10.1001/jama.2017.13836. PMID 28903154
- [Result] Elbers PW, Ince C. Mechanisms of critical illness--classifying microcirculatory flow abnormalities in distributive shock. Crit Care. 2006;10(4):221. doi: 10.1186/cc4969. PMID 16879732
- [Result] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Result] Xu JY, Ma SQ, Pan C, He HL, Cai SX, Hu SL, Liu AR, Liu L, Huang YZ, Guo FM, Yang Y, Qiu HB. A high mean arterial pressure target is associated with improved microcirculation in septic shock patients with previous hypertension: a prospective open label study. Crit Care. 2015 Mar 30;19(1):130. doi: 10.1186/s13054-015-0866-0. PMID 25887027
- [Result] Pottecher J, Deruddre S, Teboul JL, Georger JF, Laplace C, Benhamou D, Vicaut E, Duranteau J. Both passive leg raising and intravascular volume expansion improve sublingual microcirculatory perfusion in severe sepsis and septic shock patients. Intensive Care Med. 2010 Nov;36(11):1867-74. doi: 10.1007/s00134-010-1966-6. Epub 2010 Aug 20. PMID 20725823